CLINICAL TRIAL: NCT07234708
Title: Feeling Safe: Feasibility and Acceptability Study Evaluating a New Psychological Intervention for People With Psychosis and Positive Delusional Symptoms
Brief Title: Feeling Safe Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-SEG-2024-186
Record Dates: First submitted 2025-07-28; First posted 2025-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia and Schizophrenia Spectrum Psychosis
Keywords: Feeling Safe; Schizophrenia; Acceptability; Feasibility
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: Sentirnos Seguros

INTERVENTIONS:
Other: Sentirnos Seguros — The Sentirnos Seguros (Feeling Safe) programme is modular, personalised and includes the patient's preferences. The following modules are offered: improving sleep, reducing worry, increasing self-confidence, reducing the impact of voices, and feeling safe enough.

SUMMARY:
The goal of this study is to assess the acceptability and satisfaction with the psychological intervention Sentirnos Seguros (Feeling Safe) in people with psychotic disorders and positive delusional symptoms.

The main questions it aims to answer are:

* Study participants will report high levels of acceptability and satisfaction with the Sentirnos Seguros programme.
* The Sentirnos Seguros intervention will be beneficial for participants at a clinical and functional level, with higher scores in the post-treatment phase compared to the pre-treatment phase.

DETAILED DESCRIPTION:
This is a prospective, non-randomised feasibility pilot study with a before-and-after design.

The aims of the study are:

1. Assess the feasibility, acceptability, and satisfaction after receiving the Sentirnos Seguros programme in people with schizophrenia spectrum disorder and positive delusional symptoms.
2. Evaluate the clinical and functional benefits and safety of the Sentirnos Seguros programme.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and older
* Diagnosis of schizophrenia spectrum disorders and other psychotic disorders according to DSM-5
* Score ≥ 4 on the delusions item of the Positive and Negative Syndrome Scale (PANSS)
* Presence of ideas of persecution with a degree of conviction > 60% in the last 3 months

Exclusion Criteria:

* Presence of intellectual disability
* Meet DSM-5 criteria for other mental health disorders, except for substance-related and addictive disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Compliance related to the total number of successful appointments made | From baseline to 6 months (end of therapy)
  Compliance will be assessed by calculating the frequency of successful appointments from baseline to 6 months (end of therapy)
Number of drop-outs | From baseline to 6 months (end of treatment)
  The number of drop-outs will be assessed by calculating the proportion of participants who do not complete the study protocol
Acceptability, measured with an ad hoc questionnaire | From baseline to 6 months (end of the treatment)
  Acceptability with the intervention will be assessed by an ad hoc questionnaire to measure the dimensions of acceptability: perceived utility, perceived ease of use, barriers, and intention to use
Satisfaction with the intervention, measured with the Client Satisfaction Questionnaire (CSQ-8) | From baseline to 6 months (end of the treatment)
  Satisfaction with the intervention will be assessed using the CSQ-8. A 4-point Likert scale is used to rate each item (1 = very dissatisfied; 4 = very satisfied), yielding a total score ranging from 8 to 32. A low score (close to 8) indicates low satisfaction with the services received, and a high score (close to 32) indicates high satisfaction with them.

SECONDARY OUTCOMES:
Change in the severity of psychotic symptoms, measured with the Positive and Negative Syndrome Scale (PANSS) | Changes in baseline scores at 6 months
  The severity of psychotic symptoms will be assessed using the PANSS. This scale includes 30 items (7 for positive symptoms, 7 for negative symptoms, and 16 for general psychopathology). A 7-point Likert scale is used to rate each item (1 = not present; 7= most severe). The total score is the sum of all items. No specific cut-off scores have been established for the PANSS. The higher the score, the greater the clinical severity.
Change in severity of hallucinations and delusions, measured with the Psychotic Symptom Rating Scales (PSYRATS) | Changes in baseline scores at 6 months
  The severity of hallucinations and delusions will be assessed using the PSYRATS. It consists of two subscales, one for hallucinations and one for delusions, each with 17 items, with Likert-type responses ranging from 0 to 5. The final score is obtained by adding the scores for each item. It can range from 0 to 44. No specific cut-off scores have been established for the PSYRATS. The higher the score, the more severe the hallucinations/delusions.
Change in depression severity, measured with the Calgary Depresión Scale for Schizophrenia (CDSS) | Changes in baseline scores at 6 months
  The depression severity is assessed using the CDSS. This scale includes 9 items that are scored with a Likert scale that ranges from 0 (absent) to 3 (severe). The total score is the sum of all items. The higher the score, the greater the clinical severity. To identify the absence/presence of depression, a score ≥ 5 is the cut-off point.
Change in the delusional conviction severity measured with the delusional conviction-analogue visual scale (DC-VAS) | Changes in baseline scores at 6 months
  Change in the delusional conviction severity will be assessed using the DC-VAS. This scale rates the degree of conviction of the delusional idea from 0 to 10.
Change in core beliefs, measured with the Brief Core Schema Scales (BSCC) | Changes in baseline scores at 6 months
  The change in core beliefs will be assessed using the BCSS. This scale assesses an individual's core beliefs about themselves and others using a 5-point Likert scale (0-4). It comprises 24 items, yielding four scores: negative-self, positive-self, negative-others, and positive-others. Each score is based on six items. No specific cut-off scores have been established for the BCSS, scores are generally interpreted within a range. Higher scores generally indicate a greater endorsement of the beliefs represented by that subscale.
Change in safety behaviour severity, measured with the Safety Behaviour Questionnaire (SBQ) | Changes in baseline score at 6 months
  The safety behaviour severity will be assessed using the SBQ. This scale consists of 56 items rated on a 4-point Likert scale, where 0 = never and 3 = always. Specific cut-off scores haven't been established for the SBQ. Higher scores indicate greater frequency of use of safety behaviours.
Change in paranoid ideation, measured with the Spanish Green Paranoid Thought Scale (S-GPTS) | Changes in baseline scores at 6 months
  The change in paranoid ideation will be assessed using the S-GPTS. This scale consists of a total of 32 items rated on a 5-point Likert scale from 1 (Not at all) to 5 (Completely). The items are grouped into two scales of 16 items. Scale A assesses social reference ideas relevant to paranoia, while Scale B assesses persecutory thoughts. Scores on each scale range from 16 to 80 points, with higher scores reflecting a greater level of paranoid thinking. No cut-off points have been established.
Change in functioning severity, measured with the Personal and Social Performance scale (PSP) | Changes in baseline scores at 6 months
  The change in functioning severity will be assessed using the PSP scale. The PSP scale evaluates four domains: Socially Useful Activities, Personal and Social Relationships, Self-Care, and Disturbing and Aggressive Behaviours. Each domain is rated on a 6-point severity scale, which is then converted into a 10-point band score for that domain. A total score is derived from the four domain scores, resulting in a single score between 1 and 100. No cut-off score is available. Higher scores indicate better functioning across all domains, with more severe functional difficulties reflected in lower scores.
Change in self-perceived functionality severity, measured with the Self-perceived Functionality in people with Psychotic disorders (FAP-10) | Changes in baseline scores at 6 months
  The change in self-functionality will be assessed using the FAP-10. This questionnaire includes 10 items that are scored on a Likert scale ranging from 4 (Always) to 0 (Never). The total score is the sum of the scores for each item. The total score ranges from 0 (poor functionality) to 40 (excellent functionality).
Change in quality of life, measured with the Quality of Life Index (QLI-sp) | Changes in baseline scores at 6 months
  The change in quality of life will be assessed using the QLI-sp. It is a 10-item questionnaire that assesses various aspects of health-related quality of life. It is scored on a scale of 1 to 10 points, with a higher score corresponding to a better quality of life. No cut-off scores are available.
Change in recovery, measured with the Questionnaire about the Process of Recovery (QPR) | Change in baseline scores at 6 months
  The change in recovery will be assessed using the QPR. It is a 15-item scale. Each item is rated on a 5-point Likert scale, from 0 (strongly disagree) to 4 (strongly agree), and the items are added together to obtain a total recovery score. Higher scores indicate greater recovery. No cut-off scores are available.
Change in clinic insight, measured with the Scale Unawareness of Mental Disorders (SUMD) | Changes in baseline scores at 6 months
  The change in clinic insight will be assessed using the SUMD. It consists of three items that explore the degree of insight a person has into their mental disorder, the effects of medication, and the social consequences. Each item is scored from 0 to 5, where 0 indicates that the item is not relevant or cannot be assessed, and 5 indicates a lack of awareness. No cut-off points are available.
Change in cognitive insight, measured with the Beck Cognitive Insight Scale (BCIS) | Changes in baseline scores at 6 months
  The change in cognitive insight will be assessed using the BCIS. The BCIS assesses cognitive insight, specifically self-reflectiveness and self-certainty, in individuals with psychosis. It's a 15-item self-report measure where participants rate their agreement with statements on a scale of 0 to 3. The BCIS yields two subscale scores (self-reflectiveness and self-certainty) and a composite Reflectiveness-Certainty (R-C) index score. The R-C index is calculated by subtracting the self-certainty score from the self-reflectiveness score. Higher R-C index scores indicate greater cognitive insight. Cut-off scores: low cognitive insight, scores of 3 and below; moderate cognitive insight, scores of 4 to 9; and high cognitive insight, scores of 10 and above.
Presence of adverse events, measured with an ad hoc clinical interview | From baseline to 6 months (end of the intervention)
  Safety during the intervention will be assessed by collecting the presence of adverse events using an ad hoc clinical interview

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry. Hospital Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No